CLINICAL TRIAL: NCT06545656
Title: Daily Doxy: Study of Persons Receiving Daily Doxycycline to Inform Sexually Transmitted Infection Prophylaxis Regimens
Brief Title: Daily Doxycycline to Inform Sexually Transmitted Infection Prophylaxis Regimens
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Colleen Kelley, Associate Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00007429; CDC-STUDY00007429 (Other: Centers for Disease Control and Prevention)
Record Dates: First submitted 2024-08-06; First posted 2024-08-09 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Sexually Transmitted Infection
MeSH Terms: conditions — Sexually Transmitted Diseases | interventions — Doxycycline

STUDY DESIGN:
Intervention Model Description: This study aims to enroll a minimum of 10 AFAB and 10 AMAB participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Doxycycline (Experimental): Study participants taking 7 consecutive, daily doses of 100mg of Doxycycline.
  Interventions: Drug: Doxycycline

INTERVENTIONS:
Drug: Doxycycline — Doxycycline (DOX) will be given orally at 100mg doses. Participants will take the study medication for 7 consecutive days.
  Other Names: Doxy-100; Oracea; Monodox

SUMMARY:
The goal of this project is to collect data regarding the concentrations of doxycycline in mucosal tissues after daily dosing for 7 days in people assigned male sex at birth (AMAB) and assigned female sex at birth (AFAB) to inform future studies of doxycycline to protect against bacterial sexually transmitted infections (STIs).

DETAILED DESCRIPTION:
Recent studies have demonstrated the potential utility of single-dose oral doxycycline postexposure prophylaxis (Doxy-PEP) against bacterial sexually transmitted infections (STIs). Additional dosing strategies are being explored that would also provide protection from bacterial STIs. However, the pharmacokinetics of daily doxycycline and specifically the effect of this dosing on effective drug levels in mucosal tissues is underexplored. A previous pilot study conducted by the Division of human immunodeficiency virus (HIV) Prevention (DHP) Laboratory Branch at the Centers for Disease Control and Prevention (CDC) examined the ability of a single 100mg oral dose of doxycycline to penetrate the vaginal and rectal mucosa. However, data regarding daily doxycycline doses and accumulation of doxycycline with multiple doses are lacking.

The purpose of this project is to collect data regarding the ability of daily oral doxycycline taken for 7 days to concentrate in mucosal tissues in people assigned male sex at birth (AMAB) and assigned female sex at birth (AFAB). Results from this study will be compared to results of the previous pilot studies conducted by the DHP Laboratory Branch at CDC.

Healthy people assigned male or female sex at birth will take the first dose of doxycycline during the enrollment visit (Hour -144/Day -6) then will take the next 5 doses at home, one per day for the next 5 days. After 6 consecutive days of dosing, study participants will have samples collected (Hour 0/Day 0) and then will take the final dose. Rectal and vaginal swab samples will be obtained 2 to 4 hours after the final dose of doxycycline. Rectal and vaginal biopsy tissue will be collected 24 hours after the last dose.

ELIGIBILITY:
Inclusion Criteria:

* Assigned male sex or female sex at birth
* In good general health
* Not currently taking doxycycline or other tetracycline-derived antibiotics and no plans to initiate during the study
* For HIV positive people, on stable antiretroviral therapy with an undetectable viral load and cluster of differentiation 4 (CD4) count> 300ul/ml
* Willing to use condoms consistently for the duration of the study
* Able to provide informed consent
* No plans for relocation in the next 4 months
* Not pregnant and does not plan on getting pregnant for the duration of the study
* Willing to undergo peripheral blood, urine, rectal or vaginal secretion collection, and a rectal or vaginal and cervical biopsy procedure
* Willing to use study products as directed

Exclusion Criteria:

* Current or chronic history of liver disease
* Continued need for, or use during the 90 days prior to enrollment, of the following medications:

  * Systemic immunomodulatory agents
  * Supraphysiologic doses of steroids (short course steroids less than 7 days duration, allowable at the discretion of the investigators)
  * Chemotherapy or radiation for treatment of malignancy
  * Experimental medications, vaccines, or biologicals
* Intent to use doxycycline or other tetracycline-derived antibiotics during the course of the study, outside of the study procedures
* Any other clinical condition or prior therapy that, in the opinion of the investigator, would make the patient unsuitable for the study or unable to comply with the study requirements
* Known allergic reaction to study drugs
* Significant laboratory abnormalities at baseline visit for rectal biopsies, including but not limited to:

  * Hemoglobin (Hgb) ≤ 10 g/dL
  * Partial thromboplastin time (PTT) > 1.5x upper limit of normal (ULN) or international normalised ratio (INR) > 1.5x ULN
  * Platelet count <100,000

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2024-09-13 (Actual); Primary Completion 2025-04-29 (Actual); Study Completion 2025-04-29 (Actual)

PRIMARY OUTCOMES:
Doxycycline Concentration in Rectal Tissue | 24 hours after last dose (Hour 24/Day 1)
  Rectal tissue doxycycline concentrations collected 24 hours after 7 daily (T7) doses of 100 mg of doxycycline will be determined in AMAB participants.
Doxycycline Concentration in Vaginal Tissue | 24 hours after last dose (Hour 24/Day 1)
  Vaginal tissue doxycycline concentrations collected 24 hours after 7 daily (T7) doses of 100 mg of doxycycline will be determined in AFAB participants.

CONTACTS AND LOCATIONS:
Overall Officials: Colleen Kelley, MD, MPH, Principal Investigator — Emory University
Locations (1):
- Hope Clinic, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data underlie the results published for this study (including text, tables, figures, and appendices) will be made available for sharing with other researchers.
Supporting Information: Study Protocol, SAP
Time Frame: Individual participant data will be made available for sharing after publication of the primary manuscript from this study.
Access Criteria: Interested investigators can request de-identified data by email for secondary data analyses and/or meta-analyses.

DOCUMENTS (1):
  • Informed Consent Form (2025-04-16): https://cdn.clinicaltrials.gov/large-docs/56/NCT06545656/ICF_000.pdf